CLINICAL TRIAL: NCT01492725
Title: A Randomized Controlled Trial of Intra-arterial Reperfusion Therapy After Standard Dose Intravenous t-PA Within 4.5 Hours of Stroke Onset Utilizing Dual Target Imaging Selection.
Brief Title: Extending the Time for Thrombolysis in Emergency Neurological Deficits - Intra-Arterial
Acronym: EXTEND-IA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: On DSMB advice, trial recruitment has been halted for efficacy. F/U continues
Sponsor: Neuroscience Trials Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTA1101
Record Dates: First submitted 2011-11-20; First posted 2011-12-15 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2014-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-arterial Clot Retrieval after iv tPA (Experimental)
  Interventions: Device: Intra-arterial Clot Retrieval with Solitaire device
- Standard care iv tPA (Active Comparator)
  Interventions: Genetic: intravenous tissue plasminogen activator (tPA)

INTERVENTIONS:
Device: Intra-arterial Clot Retrieval with Solitaire device — Intra-arterial mechanical clot retrieval with the Solitaire device after patients have received standard therapy with intravenous tissue plasminogen activator (tPA). Clot retrieval involves cerebral angiography and takes approximately 2 hours.
  Arms: Intra-arterial Clot Retrieval after iv tPA
Genetic: intravenous tissue plasminogen activator (tPA) — Standard care IV tPA therapy administered as per registered product information
  Arms: Standard care iv tPA

SUMMARY:
Patients presenting to the emergency department with acute ischaemic stroke, who are eligible for standard intravenous tPA therapy within 4.5 hours of stroke onset will be assessed for "dual target" major vessel occlusion and mismatch to determine their eligibility for randomisation into the trial. If the patient gives informed consent they will be randomised 50:50 using central computerised allocation to intra-arterial clot retrieval after IV tPA or IV tPA alone. The trial is prospective, randomised, open-label, blinded endpoint (PROBE) design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with anterior circulation acute ischaemic stroke eligible using standard criteria to receive IV tPA within 4.5 hours of stroke onset
2. Patient, family member or legally responsible person depending on local ethics requirements has given informed consent
3. Patient"s age is ≥18 years
4. Intra-arterial clot retrieval treatment can commence (groin puncture) within 6 hours of stroke onset.

   Imaging inclusion criteria

   Dual target:
5. Arterial occlusion on CTA or MRA of the ICA, M1 or M2
6. Mismatch - Using CT or MRI with a Tmax >6 second delay perfusion volume and either CT-rCBF or DWI infarct core volume. a) Mismatch ratio of greater than 1.2, and b) Absolute mismatch volume of greater than 10 ml, and. c) Infarct core lesion volume of less than 70mL

Exclusion Criteria:

1. Intracranial haemorrhage (ICH) identified by CT or MRI
2. Rapidly improving symptoms at the discretion of the investigator
3. Pre-stroke mRS score of ≥ 2 (indicating previous disability)
4. Inability to access the cerebral vasculature in the opinion of the neurointerventional team
5. Contra indication to imaging with MR with contrast agents
6. Participation in any investigational study in the previous 30 days
7. Any terminal illness such that patient would not be expected to survive more than 1 year
8. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
9. Pregnant women
10. Previous stroke within last three months
11. Recent past history or clinical presentation of ICH, subarachnoid haemorrhage (SAH), arterio-venous (AV) malformation, aneurysm, or cerebral neoplasm. At the discretion of each Investigator.
12. Current use of oral anticoagulants and a prolonged prothrombin time (INR > 1.6)
13. Use of heparin, except for low dose subcutaneous heparin, in the previous 48 hours and a prolonged activated partial thromboplastin time exceeding the upper limit of the local laboratory normal range.
14. Use of glycoprotein IIb - IIIa inhibitors within the past 72 hours. Prior use of single or dual agent oral platelet inhibitors (clopidogrel and/or low-dose aspirin) is permitted.
15. Clinically significant hypoglycaemia.
16. Uncontrolled hypertension defined by a blood pressure > 185 mmHg systolic or >110 mmHg diastolic on at least 2 separate occasions at least 10 minutes apart, or requiring aggressive treatment to reduce the blood pressure to within these limits. The definition of "aggressive treatment" is left to the discretion of the responsible Investigator.
17. Hereditary or acquired haemorrhagic diathesis
18. Gastrointestinal or urinary bleeding within the preceding 21 days
19. Major surgery within the preceding 14 days which poses risk in the opinion of the investigator.
20. Exposure to a thrombolytic agent within the previous 72 hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reperfusion at 24 hours (CT or MR perfusion imaging) | 24 hours post stroke onset
Favourable clinical response at 3 days(National Institutes of Health Stroke Score - NIHSS) | 3 days post stroke onset
  NIHSS - reduction >/= 8 points or reaching 0-1)

SECONDARY OUTCOMES:
Reperfusion at 24 hrs post stroke without symptomatic intracerebral hemorrhage (CT or MR perfusion imaging) | 24 hours post stroke onset
Recanalisation at 24 hrs post stroke (CT or MR angiography) | 24 hours post stroke onset
Infarct growth within 24 hrs (CT and MRI) | 24 hours post stroke onset
Stroke severity (NIHSS) at 24 hours | 24 hours post stroke onset
Symptomatic intra-cranial hemorrhage (ECASS type 2 parenchymal hematoma on CT or MRI combined with >/=4 point deterioration in NIHSS within 36 hours of treatment). | within 36 hours of intervention
Death due to any cause | 3 months
Modified Rankin Scale (mRS) 0-1 at 3 months | 3 months
Categorical shift in mRS at 3 months | 3 months
NIHSS reduction 8 points or reaching 0-1 at 3 months | 3 months
Modified Rankin Scale (mRS) 0-2 at 3 months | 3 months

CONTACTS AND LOCATIONS:
Locations (9):
- Australia (8):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Western Hospital, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- Auckland Hospital, Grafton, Auckland, New Zealand

REFERENCES:
- [Derived] Sarraj A, Albers GW, Mitchell PJ, Hassan AE, Abraham MG, Blackburn S, Sharma G, Yassi N, Kleinig TJ, Shah DG, Wu TY, Hussain MS, Tekle WG, Gutierrez SO, Aghaebrahim AN, Haussen DC, Toth G, Pujara D, Budzik RF, Hicks W, Vora N, Edgell RC, Slavin S, Lechtenberg CG, Maali L, Qureshi A, Rosterman L, Abdulrazzak MA, AlMaghrabi T, Shaker F, Mir O, Arora A, Martin-Schild S, Sitton CW, Churilov L, Gupta R, Lansberg MG, Nogueira RG, Grotta JC, Donnan GA, Davis SM, Campbell BCV; SELECT, EXTEND-IA, EXTEND-IA TNK, and EXTEND-IA TNK Part-II Investigators. Thrombectomy Outcomes With General vs Nongeneral Anesthesia: A Pooled Patient-Level Analysis From the EXTEND-IA Trials and SELECT Study. Neurology. 2023 Jan 17;100(3):e336-e347. doi: 10.1212/WNL.0000000000201384. Epub 2022 Oct 26. PMID 36289001
- [Derived] Ng FC, Churilov L, Yassi N, Kleinig TJ, Thijs V, Wu T, Shah D, Dewey H, Sharma G, Desmond P, Yan B, Parsons M, Donnan G, Davis S, Mitchell P, Campbell B. Prevalence and Significance of Impaired Microvascular Tissue Reperfusion Despite Macrovascular Angiographic Reperfusion (No-Reflow). Neurology. 2022 Feb 22;98(8):e790-e801. doi: 10.1212/WNL.0000000000013210. Epub 2021 Dec 14. PMID 34906976
- [Derived] Campbell BCV, Mitchell PJ, Churilov L, Keshtkaran M, Hong KS, Kleinig TJ, Dewey HM, Yassi N, Yan B, Dowling RJ, Parsons MW, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Rice H, de Villiers L, Ma H, Desmond PM, Meretoja A, Cadilhac DA, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular Thrombectomy for Ischemic Stroke Increases Disability-Free Survival, Quality of Life, and Life Expectancy and Reduces Cost. Front Neurol. 2017 Dec 14;8:657. doi: 10.3389/fneur.2017.00657. eCollection 2017. PMID 29312109
- [Derived] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Derived] Campbell BC, Mitchell PJ, Yan B, Parsons MW, Christensen S, Churilov L, Dowling RJ, Dewey H, Brooks M, Miteff F, Levi C, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Kleinig T, Scroop R, Chryssidis S, Barber A, Hope A, Moriarty M, McGuinness B, Wong AA, Coulthard A, Wijeratne T, Lee A, Jannes J, Leyden J, Phan TG, Chong W, Holt ME, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA investigators. A multicenter, randomized, controlled study to investigate EXtending the time for Thrombolysis in Emergency Neurological Deficits with Intra-Arterial therapy (EXTEND-IA). Int J Stroke. 2014 Jan;9(1):126-32. doi: 10.1111/ijs.12206. Epub 2013 Nov 10. PMID 24207098